CLINICAL TRIAL: NCT04263012
Title: Establishment of a LVAD Destination Program in a Swiss Non Cardiac Transplant University Hospital: 5 Year Experience
Brief Title: Establishment of a LVAD Destination Program in a Swiss Non Cardiac Transplant University Hospital
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00017; ch19Grapow2
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Heart Implant Complication
Keywords: left ventricular assist device (LVAD); heart; implant; artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with an implanted LVAD: Patients which received an implantation of a left ventricular assist device (LVAD) at the University Hospital Basel since 2014
  Interventions: Other: collection of patient data

INTERVENTIONS:
Other: collection of patient data — assess mortality rate, rehospitalization and survival rate of patients after receiving an artificial heart implant

SUMMARY:
The goal of this study is to demonstrate the challenges and the effort to set up an artificial heart program as well as to report about the follow-up treatment and the mortality rate

ELIGIBILITY:
Inclusion Criteria:

* Patients who received an LVAD implant

Exclusion Criteria:

* not enough data collected
* stated will of the Patient, that his data can not be used

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who received an LVAD implant
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
30 days mortality | 30 days after surgery
  mortality rate 30 days after receiving the LVAD implant
rehospitalization rate | between day of surgery and 31.12.2019
  rehospitalization rate of patients after receiving the LVAD implant

SECONDARY OUTCOMES:
survival rate | between day of surgery and 31.12.2019
  survival rate of patients after receiving the LVAD implant (Kaplan-Meier curve)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Grapow, Prof Dr. med., Principal Investigator — Herzzentrum Hirslanden Zürich
Locations (1):
- Herzchirurgie University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Schaeffer T, Pfister O, Mork C, Mohacsi P, Rueter F, Scheifele S, Morgen A, Zenklusen U, Doebele T, Maurer M, Erb J, Fassl J, Cueni N, Siegemund M, Pargger H, Gahl B, Osswald S, Eckstein F, Grapow M. 5-year results of a newly implemented mechanical circulatory support program for terminal heart failure patients in a Swiss non-cardiac transplant university hospital. J Cardiothorac Surg. 2021 Mar 31;16(1):64. doi: 10.1186/s13019-021-01447-5. PMID 33789723